CLINICAL TRIAL: NCT05443360
Title: A Randomized, Double-blind, Active-controlled Study to Evaluate the Effects of Amorphous Calcium Carbonate in Rheumatoid Arthritis Patients With Osteopenia or Osteoporosis
Brief Title: To Evaluate the Efficacy and Safety of Amorphous Calcium Carbonate in RA Patient With Osteopenia or Osteoporosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Der-Yuan Chen, Rheumatology and Immunology Center, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CMUH111-REC2-014
Record Dates: First submitted 2022-06-15; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Rheumatoid Arthritis; Osteopenia or Osteoporosis
MeSH Terms: conditions — Arthritis, Rheumatoid; Bone Diseases, Metabolic; Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- amorphous calcium carbonate (ACC group) (Experimental): oral use, 2 ACC tablets (1000 mg / tablet, 200 mg calcium element / tablet) twice daily given after breakfast and dinner.
  Interventions: Dietary Supplement: DENSITY™ (Amorphous calcium carbonate, ACC)
- crystalized calcium carbonate (CCC group) (Active Comparator): oral use, 2 CCC tablets (1000 mg / tablet, 200 mg calcium element / tablet) twice daily given after breakfast and dinner.
  Interventions: Dietary Supplement: Crystalized calcium carbonate (CCC)

INTERVENTIONS:
Dietary Supplement: DENSITY™ (Amorphous calcium carbonate, ACC) — 1. Dosage form: tablet
  2. Dose(s): 1000 mg /tablet, comprising 500 mg amorphous calcium carbonate per tablet (calcium element 200mg)
  3. Dosing schedule: The usual dose for oral use is 2 ACC tablets (400 mg calcium element) twice daily given after breakfast and dinner.
  Arms: amorphous calcium carbonate (ACC group)
Dietary Supplement: Crystalized calcium carbonate (CCC) — 1. Dosage form: tablet
  2. Dose(s): 1000 mg /tablet, comprising 500 mg crystalized calcium carbonate per tablet (calcium element 200mg)
  3. Dosing schedule: The usual dose for oral use is 2 CCC tablets (400 mg calcium element) twice daily given after breakfast and dinner.
  Arms: crystalized calcium carbonate (CCC group)

SUMMARY:
DensityTM, an amorphous calcium carbonate (ACC) imported by Universal Integrated Corporation, is tried to demonstrate its efficacy and safety in rheumatoid arthritis patient with osteopenia or osteoporosis, compared to crystalized calcium carbonate (CCC).

DETAILED DESCRIPTION:
This is a randomized, double-blind, active-controlled study to evaluate the efficacy and safety of amorphous calcium carbonate in rheumatoid arthritis patients with osteopenia or osteoporosis, compared to crystalized calcium carbonate.

A total of 180 subjects will be enrolled into this study. Eligible subjects will be randomized to receive amorphous calcium carbonate (ACC group) or crystalized calcium carbonate (CCC group) with 1:1 allocation. Randomization will be stratified by the use of biologics. The study product, 2 tablets (400mg calcium element), will be taken twice daily approximately 30 minutes after breakfast and dinner during 12-month treatment period. Additional 600 IU vitamin D3 will be also received with investigational product after breakfast.

The study will consist of 7 clinical visits. Subjects will come to the clinics at Visit 1 (screening visit), Visit 2 (randomization, regimen start), Visit 3 to 6 (follow-up visits), and Visit 7 (post-treatment follow-up visits) according to the pre-defined schedule.

The DXA score, and BTM (P1NP, CTX) from fasting serum samples, and FRAX score will be collected. The treatment-emergent adverse events for safety endpoints will be also recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≧45 years of age.
2. Diagnosis of rheumatoid arthritis according to 2010 American College of Rheumatology Guideline (ACR Guideline), with severe osteopenia or osteoporosis.
3. With a DAS28 (Disease Activity Score 28) score ranged from 2.6 to 5.1 at screening visit.
4. With a documented DXA score ≦-2.0 at the lumbar spine or total hip and without compression fracture within the 3 months prior to screening visit.
5. With a FRAX score at least medium risk (major osteoporotic fracture 10-19%, hip fracture 1-3%) at screening visit.
6. Willingness to limit additional vitamin D3 intake to 600 IU per day during the study period.
7. Ability to complete the entire procedure and to comply with study instructions.
8. Will provide completed and signed written informed consents.

Exclusion Criteria:

1. History of or current diseases that may interfere serum calcium, such as hypocalcemia, hypercalcemia, hyperparathyroidism, hypoparathyroidism, hyperthyroidism or hypothyroidism, or other metabolic bone disease, from any cause within 1 year prior to screening.
2. Chronic kidney disease with receiving peritoneal dialysis or hemodialysis
3. Known hypersensitivity to any component of the study product.
4. Current treatment with any anti-osteoporotic drug (i.e. bisphosphonates, Denosumab (Prolia), teriparatide (Forteo), Romosozumab (Evenity), Raloxifene (Evista), etc.).
5. Any previous or ongoing clinically significant illness that may interfere with the study conduct, as judged by the investigator.
6. Participation in any other investigational study within 30 days prior to receiving study medication.
7. Any condition that in the opinion of the investigator would jeopardize the evaluation of efficacy or safety.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in bone mineral density (BMD) measured by dual-energy x-ray absorptiometry (DXA) in lumbar spine and total hip at Month 13 | 12 months
  The BMD and the corresponding change from baseline will be summarized with descriptive statistics and the 95% CI by study groups. The difference in mean change from baseline in BMD between study groups will be analyzed by two sample t test. Additionally, the intra-group difference will be analyzed by paired t test.

SECONDARY OUTCOMES:
Percentage change from baseline in bone mineral density (BMD) measured by dual-energy x-ray absorptiometry (DXA) in lumbar spine and total hip at Month 13 | 12 months
  The percentage change from baseline in BMD measured by DXA in lumbar spine and total hip at Month 13 will be summarized with descriptive statistics and the 95% CI by study groups. The difference in percentage change from baseline in BMD between study groups will be analyzed by two sample t test.
Responder number and rate in bone mineral density (BMD) measured by dual-energy x-ray absorptiometry (DXA) in lumbar spine and total hip at Month 13 | 12 months
  The responder is defined as 20% reduction in DXA score from the baseline. The responder will be presented as count and percentage in frequency table, and the 95% exact (Clopper-Pearson) CI will be provided as well by study group. Fisher's exact test will be used for the comparison between study groups.
FRAX score (Fracture Risk Assessment Tool) change from baseline at Visit 1, 4, and 6 | 12 months
  The FRAX score and the corresponding change from baseline at Visit 1, 4, and 6 will be summarized with descriptive statistics and the 95% CI by study groups. The difference in mean change from baseline in FRAX score between study groups will be analyzed by two sample t test. Additionally, the intra-group difference will be analyzed by paired t test.
Bone turnover markers (BTM) change from baseline level 5.1 P1NP (total procollagen type 1 N-terminal propeptide) 5.2 CTX (C-terminal telopeptide of type 1 collagen) | 12 months
  The bone turnover markers (BTM) includes P1NP (total procollagen type 1 N-terminal propeptide) and CTX (C-terminal telopeptide of type 1 collagen). For the bone turnover markers (BTM), the descriptive summary of original values and the change from baseline will be provided by study groups. Two sample t test will be used for the comparison of study groups in change from baseline be. Additionally, the intra-group comparison will be analyzed by paired t test.

CONTACTS AND LOCATIONS:
Overall Officials: Der-Yuan Chen, Doctor, Principal Investigator — Rheumatology and Immunology Center; Wei-Sheng Chen, Doctor, Principal Investigator — Division of Allergy, immunology and Rheumatology
Locations (2):
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei